CLINICAL TRIAL: NCT01961791
Title: Lymph Node Staging System With a Novel Concept for Gastric Cancer: a Hybrid Type of Topographic and Numeric Ones
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2012-0798
Record Dates: First submitted 2013-10-09; First posted 2013-10-11 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Gastrectomy for Gastric Cancer
Keywords: gastric cancer, staging system, prognosis
MeSH Terms: conditions — Stomach Neoplasms | interventions — Gastrectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TNM 7th edition: staged by the current TNM 7th edition of AJCC/UICC
  Interventions: Procedure: gastrectomy
- new TNM stage: staged by new TNM stage with new lymph node staging concept
  Interventions: Procedure: gastrectomy

INTERVENTIONS:
Procedure: gastrectomy — gastrectomy with D1 + lymph node dissection for clinically early gastric cancer, and gastrectomy with D2 lymph node dissection for clinically advanced gastric cancer

SUMMARY:
For staging the status of lymph node metastasis in gastric cancer, typographic based staging system was applied until last decade, especially in Eastern countries. However the old typographic lymph node staging system in gastric cancer was too complicated and less accurate for predicting the prognosis. Now the numeric based lymph node staging system is used in both East and West, but it include problems: no information on the anatomical extent of the disease, preoperative lymph node staging is nearly impossible, failure to provide an appropriate treatment plan, cannot represent the extent of lymph node dissection. We designed simple and specifically representing the anatomic extent of the disease for staging the status of lymph node in gastric cancer. Thus we compared its prognostic performance of this new staging system with those of the current TNM 7th edition of AJCC/UICC.

ELIGIBILITY:
Inclusion Criteria:

* patients were pathologically confirmed as primary gastric cancer
* patients underwent gastrectomy with curative intent.

Exclusion Criteria:

* Patients underwent minimally invasive surgery
* patients with any distant metastases including peritoneal seeding and para-aortic LNs metastasis)
* when the location of lymph nodes were not divided
* patients underwent chemotherapy preoperatively
* patients had metastatic lymph nodes with unclear location

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent gastrectomy with lymph node dissection for gastric cancer in Yonsei University Hospital, Seoul
Sampling Method: Non-Probability Sample
Enrollment: 6025 (Actual)
Dates: Start 2000-01; Primary Completion 2011-12 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Prognostic performance | participants will be followed for the duration of survival, an expected average of 36 months.
  The overall survival (OS) was used to evaluate the prognosis after gastrectomy. The Kaplan-Meier method and log-rank test were applied to analyze the OS. In addition, the Cox proportional hazards model was used to estimate hazard ratios (HRs). To compare the discrimination of each stage, the Kaplan-Meier curves from each stage in both staging systems was used. For comparing prognostic performance of each staging system, Harrell C-index (for measuring the predictive accuracy of survival outcome) were used.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Crew KD, Neugut AI. Epidemiology of gastric cancer. World J Gastroenterol. 2006 Jan 21;12(3):354-62. doi: 10.3748/wjg.v12.i3.354. PMID 16489633
- [Background] Brierley JD, Catton PA, O'Sullivan B, Dancey JE, Dowling AJ, Irish JC, McGowan TS, Sturgeon JF, Swallow CJ, Rodrigues GB, Panzarella T. Accuracy of recorded tumor, node, and metastasis stage in a comprehensive cancer center. J Clin Oncol. 2002 Jan 15;20(2):413-9. doi: 10.1200/JCO.2002.20.2.413. PMID 11786568
- [Background] Karpeh MS, Leon L, Klimstra D, Brennan MF. Lymph node staging in gastric cancer: is location more important than Number? An analysis of 1,038 patients. Ann Surg. 2000 Sep;232(3):362-71. doi: 10.1097/00000658-200009000-00008. PMID 10973386
- [Background] Sayegh ME, Sano T, Dexter S, Katai H, Fukagawa T, Sasako M. TNM and Japanese staging systems for gastric cancer: how do they coexist? Gastric Cancer. 2004;7(3):140-8. doi: 10.1007/s10120-004-0282-7. PMID 15449201
- [Background] Fujii K, Isozaki H, Okajima K, Nomura E, Niki M, Sako S, Izumi N, Mabuchi H, Nishiguchi K, Tanigawa N. Clinical evaluation of lymph node metastasis in gastric cancer defined by the fifth edition of the TNM classification in comparison with the Japanese system. Br J Surg. 1999 May;86(5):685-9. doi: 10.1046/j.1365-2168.1999.01115.x. PMID 10361195